CLINICAL TRIAL: NCT05612438
Title: RADIX 2 RENAL ARTERY STENT Evaluation of Safety and Performance in Everyday Clinical Practice: Post-Market Retrospective Study.
Brief Title: RADIX 2 RENAL STENT Post-Market Retrospective Study
Acronym: RADIX 2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CID S.p.A. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: P12204
Record Dates: First submitted 2022-11-04; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Renal Artery Stenosis; Renal Failure
MeSH Terms: conditions — Renal Artery Obstruction; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RADIX 2 Stent — RADIX 2 stent implantation for the treatment of occlusive lesions of the native renal arteries; or in the case of inadequate results (residual stenosis > 30%) or dissection of the vessel wall following PTRA procedure with or without stenting.

SUMMARY:
The Carbostent™ Radix 2 stent is a CE marked balloon expandable bare metal stent for the treatment of renal artery stenosis.

The aim of this post-market retrospective study protocol P12204, is to collect clinical data on patients treated with the RADIX 2 stent in routine clinical practice.

In order to obtain long-term follow-up data, the data collection will be limited to patients that have been treated with the Radix 2 stent at least 12 months prior to the study start.

DETAILED DESCRIPTION:
The objective of this post-market study is collect retrospective clinical data on the implantable medical device Radix 2 stent in an unselected population treated in the current clinical practice. Data will be collected via medical chart review in anonymous form.

Radix2 is a bare metal balloon expandable stent with a progressive multicellular design for treatment of renal artery stenosis. The stent is stent coated with i-Carbofilm™ to accelerate the rate of endothelization and strut coverage.

The product is CE marked and commercially available since July 2010. Additional technical information on RADIX2 is available online: http://www.alvimedica.com/Product/15/bms-b-e-radix2

ELIGIBILITY:
Inclusion Criteria:

The study will be conducted in the "real world" population, according to the following criteria.

Selection criteria:

* Patient has been implanted with at least one study stent (Radix2) according to the indications described in the IFU.
* Study Device Implanted is at least12 months prior to the starting date of the retrospective anonymous data collection.

Exclusion Criteria:

* Patients treated less than 12 months prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected with occlusive lesions of the native renal artery disease treated with the study stent, these patients are generally affected by cardiovascular comorbidities with a high incidence of mortality or in the terminal phase of the disease or in advanced age and in serious health conditions
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-03 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Major renal events | 30 days
  Major renal events at 30 days - composite of:
  death from renal causes, related to study device or procedure; embolic events related to study device or procedure, resulting in kidney damage; acute kidney injury Stage 3 (AKIN criteria); ipsilateral nephrectomy, related to the study device or procedure.

SECONDARY OUTCOMES:
Acute device success | 24 hours
  Acute Device Success, defined as the successful delivery of the assigned device(s) to the designated target location
Technical success | 24 hours
  Technical Success, defined as the ability to implant the stent with a residual angiographic stenosis no greater than 30%
In Stent Restenosis | 12 months
  Restenosis of Radix2 stent, requiring repeat revascularization
Arterial Blood Pressure | 12 months
  Systolic and diastolic arterial blood pressure changes during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeller T, Rastan A, Kliem M, Schwarzwalder U, Frank U, Burgelin K, Schwarz T, Amantea P, Muller C, Neumann FJ. Impact of carbon coating on the restenosis rate after stenting of atherosclerotic renal artery stenosis. J Endovasc Ther. 2005 Oct;12(5):605-11. doi: 10.1583/05-1599MR.1. PMID 16212462
- See also: Manufacturer website — http://www.alvimedica.com/
- See also: Clinical Research Organization — https://meditrial.net/